CLINICAL TRIAL: NCT03411837
Title: Dupilumab Registry Study
Brief Title: Dupilumab Phase 4 Study
Acronym: DRS
Status: Terminated | Type: Observational
Why Stopped: Investigator moved from institution.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jonathan Silverberg, MD, PhD, MPH, Northwestern University
Other Study IDs: STU00088226
Record Dates: First submitted 2017-11-13; First posted 2018-01-26 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis, dupilumab
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dupilumab: Patients with moderated-to-severe atopic dermatitis who are receiving dupilumab as a standard of care
  Interventions: Biological: Dupilumab

INTERVENTIONS:
Biological: Dupilumab — Biologic (monoclonal antibody)
  Other Names: Dupixent

SUMMARY:
The investigators will monitor for the incidence of adverse-events in a prospective, longitudinal, non-interventional and observational real-world sub-study of adults patients with moderate-to-severe AD who are receiving dupilumab as standard-of-care therapy.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, longitudinal, non-interventional and observational sub-study of patients receiving dupilumab as normal standard-of-care treatment to assess the efficacy (Specific Aim #1) and safety (Specific Aim #2) of dupilumab for the treatment of moderate-to-severe AD, as well as the prevention and/or mitigation of comorbid health conditions (Specific Aim #3). This study will address the hypotheses that dupilumab will lead to improved long-term control and decreased severity of AD, and that long-term monitoring will shed light on the incidence of adverse drug events.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over who have been diagnosed with Atopic Dermatitis and are using dupilumab therapy as part of standard of care.
* Parents of adolescents ages 12 to 17 who have been diagnosed with Atopic Dermatitis and are receiving dupilumab off-label for the management of AD.

Exclusion Criteria:

* Patients not on dupilumab
* Those who do not comply with the study requirements
* Those who do not provide informed consent

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with moderate-to-severe atopic dermatitis on dupilumab
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Quantified Itch Survey | 1 to 3 months
Quantified Sleep Survey | 1 to 3 months
Quantified Quality of Life Survey | 1 to 3 months

SECONDARY OUTCOMES:
Occurrence of any AEs by 24 months | 24 months
  Will be determined based off of patient reported safety events
Occurrence of any infections by 24 months | 24 months
  Will be determined based off of patient reported safety events
Occurrence of any SAEs by 24 months | 24 months
  Will be determined based off of patient reported safety events

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States